## Post Extraction Wound Healing Evaluation of Immediate Complete Denture using IPR Scale

[NCT ID not yet assigned]

Unique Protocol ID: 01154777474

**Document Date: 15/7/2022** 

## **Assessment and Treatment Planning**

All patients should have a thorough history, clinical examination and any relevant investigations carried out to attain a correct diagnosis and treatment plan.

The formulated diagnoses and treatment plan as well as the costs and timeframes involved need to be thoroughly discussed with the patient to obtain informed consent before proceeding with treatment. It is also vital that the clinician has a clear understanding of the patient's expectations of treatment and whether these can be achieved in the proposed treatment, particularly in those patients who have never worn dentures before. Patients need to be clearly made aware of the limitations of a removable prosthesis in general and also the issues associated with an immediate denture. Denture wearing is a complex phenomenon and while the technical ability of the clinician has a huge role to play in its success, it is largely dependent on the patient's psychological acceptance and neuromuscular ability to cope with the dentures.